CLINICAL TRIAL: NCT05750173
Title: Pre-procedural Assessment of Coronary Artery Disease in Patients Undergoing Transcatheter Aortic Valve Implantation (TAVI) - Comparision of Pre-TAVI CTA vs. Pre-TAVI ICA
Brief Title: The EASE-IT CT Registry
Status: Recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: EASE-IT CT
Record Dates: First submitted 2022-12-08; First posted 2023-03-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Transcatheter Aortic Valve Implantation (TAVI)
Keywords: TAVI; Transcatheter Aortic Valve Implantation; severe Aortic Stenosis; sAS; computed tomography angiography; CTA; invasive coronary angiography; ICA; Coronary Artery Disease; CAD
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Investigational CTA-only cohort: 100 consecutive patients that are not already diagnosed with significant (≥50%) proximal stenosis of the left anterior descending artery (LAD) OR the left main coronary artery (LM) and who have not previously undergone coronary revascularisation.
  Interventions: Other: Streamlining of the pre-procedural patient pathway
- CTA+ICA control cohort: At least 50 consecutive patients who have not already been diagnosed with significant (≥50%) LM / proximal LAD stenosis an who have not previously undergone conronary revascularisation and will undergo CTA. If LM / proximal LAD stenosis of ≥50% can be ruled out and ICA is also performed prior to TAVI these patients will serve as control group.
  Interventions: Other: Streamlining of the pre-procedural patient pathway

INTERVENTIONS:
Other: Streamlining of the pre-procedural patient pathway — Pre-TAVI ICA is associated with procedural risk, radiation, costs and requires hospitalization (2d).
  Show that CTA is a viable alternative to rule out ≥50% left main coronary artery (LM) / prox. left anterior descending artery (LAD) stenosis.
  An implementation of a standardized patient pathway which is reproducible, will help to streamline the pre-procedural workup of patients without compromising patient safety.

SUMMARY:
ICA is not always required for a pre-TAVI workup of octogenarians and can be substituted by CTA resulting in a streamlined pre-procedural workup of patients without compromising patient safety.

DETAILED DESCRIPTION:
Patients undergoing TAVI require routine pre-procedural assessment of CAD (coronary artery disease).

ICA (invasive coronary angiography) is the gold standard in patients with high pre-test probability. It is associated, however, with procedural risk, radiation and cost.

CTA (computed tomography angiography) currently has limited use for the evaluation of CAD in pts with severe symptomatic AS (aortic stenosis) - medications required such as beta blockers and nitroglycerine, are frequently not well tolerated by pts.

But as TAVI is increasingly being performed in patients with modest pre-test probabilities for obstructive CAD or a lack of implications thereof (pts. ≥75 yrs), the use of CTA may become more appealing.

ELIGIBILITY:
Inclusion Criteria:

Investigational CTA-only Cohort

* Consecutive adult patients ≥ 75 years
* Consecutive patients with severe AS (symptomatic or asymptomatic) with a guideline-based indication to undergo implantation of a transcatheter heart valve of the SAPIEN family
* Ability to undergo CTA
* Patient is scheduled to undergo a 30 Day and 3 Months follow-up

CTA+ICA control Cohort

* Consecutive adult patients ≥ 75 years
* Consecutive patients underwent implantation of a transcatheter heart valve of the SAPIEN family because of severe aortic stenosis
* Ability to undergo CTA and ICA

Exclusion Criteria:

investigational CTA-only Cohort

* Patients with already diagnosed proximal stenosis of the left anterior descending artery (LAD) OR the left main coronary artery (LM) ≥50%
* Any prior coronary revascularization / prior aortic valve replacement
* Life expectancy below 12 months
* Lack of informed consent / data protection statement

CTA+ICA control Cohort

* Patients diagnosed with proximal stenosis of the left anterior descending artery (LAD) OR the left main coronary artery (LM) ≥50% already at baseline
* Any prior coronary revascularization / prior aortic valve replacement
* Life expectancy below 12 months
* Lack of informed consent / data protection statement

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Investigational CTA-only phase:
  100 consecutive patient who have not already been diagnosed with significant (≥50%) left main coronary artery (LM) or proximal stenosis of the left anterior descending artery (LAD) ans who have not previously undergone coronary revascularisation.
  CTA+ICA control phase:
  50 consecutive patients who have not alreeady been diagnosed with significant (≥50%) left main coronary artery (LM) / proximal LAD stenosis and who have not previously undergone coronary revascularisation and will undergo CTA. If LM/ proximal LAD stenosis of (≥50%) can be ruled out and ICA is also performed prior to TAVI these patients will serve as control group.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Number and percentage of patients experiencing CAD specific outcomes in each group at 30 days after TAVI | 30 days
  CAD specific combined "endpoint" at 30 days
  * All-cause death
  * Non-fatal myocardial infarction
  * Ischemia-driven revascularization
  * Rehospitalization (valve- or procedure-related including heart failure)
  * Life-threatening/disabling or major bleeding
  Number and percentage of subjects with above specified outcomes at 30 days
Comparison of the Number and percentage of patients experiencing CAD specific outcomes in each group at 3 months after TAVI | 3 months
  CAD specific combined "endpoint" at 3 months
  * All-cause death
  * Non-fatal myocardial infarction
  * Ischemia-driven revascularization
  * Rehospitalization (valve- or procedure-related including heart failure)
  * Life-threatening/disabling or major bleeding
  Number and percentage of subjects with above specified outcomes at 3 months.
Number and percentage of patients with Device success assessed at 30 days after TAVI using the VARC3 criteria | 30 days
  VARC-3 defined device success at 30 days:
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation)
  Number and percentage of subjects with device success at 30 days as per VARC-3 definition.
Number and percentage of patients free from Device safety issues assessed at 30 days after TAVI using the VARC3 criteria | 30 days
  VARC-3 defined early safety at 30 days:
  * Freedom from all-cause mortality
  * Freedom from all Stroke
  * Freedom from all VARC type 2-4 bleeding
  * Freedom from all major vascular, access-related, or cardiac structural complication
  * Freedom from all acute kidney injury stage III/IV
  * Freedom from all moderate/severe aortic regurgitation
  * Freedom from all new permanent pacemaker implantations due to procedure-related conduction abnormalities
  * Freedom from all surgery/intervention related to the device
  Number and percentage of subjects free from VARC3-defined safety issues at 30 days as per VARC-3 definition.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mascherbauer, Prof. Dr., Principal Investigator — Clinical Department for Internal Medicine 3, University Hospital St. Pölten, Austria
Locations (6):
- Austria (4):
  - Universitätsklinik für Innere Medizin III - Kardiologie und Angiologie, Innsbruck, Tyrol
  - University Clinic St. Pölten, Sankt Pölten
  - Medical University of Vienna, Vienna
  - Klinik Floridsdorf, Vienna
- Germany (2):
  - University Hospital Bochum / HDZ NRW, Bad Oeynhausen, North Rhine-Westphalia
  - University Hospital of the Bergmannsheil gGmbH, Bochum, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No
no individual participant data (IPD) will be shared